CLINICAL TRIAL: NCT02239133
Title: Pilot Study for the Evaluation of the ProVATE (ProTIPI) Pessary Designs in the Temporary Management of Pelvic Organ Prolapse (POP) in Women
Brief Title: R&D Supporting Pilot Study for the Assessment of the Safety and Effectiveness of the ProVATE (ProTIPI) Vaginal Pessary
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ConTIPI Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProVATE PT 103
Record Dates: First submitted 2014-09-08; First posted 2014-09-12 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; POP
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ProVATE vaginal pessary (Experimental): The ProVATE device is a disposable, single-use, vaginal pessary for the management of Pelvic Organ Prolapse ("POP"). The ProVATE device is similar to other ring pessaries currently on the market. Its features allow for easy and comfortable insertion and removal by the user herself at her home environment. The ProVATE device is provided in six (6) different sizes and is intended for prescription use only.
  Interventions: Device: ProVATE vaginal pessary

INTERVENTIONS:
Device: ProVATE vaginal pessary

SUMMARY:
The study includes five (5) main stages: Screening, Enrollment, Size fitting, Usage and Termination.

Subject screening will be held during visit one (1) and visit two (2) at the clinic.

Initiation and Size fitting:

All eligible subjects will undergo size fitting by a gynecologist / urogynecologist, during visit 2, to find the suitable size for her. The subject will use the ProVATE device of the chosen size at the clinic vicinity for about one (1) hour and for 40-80 hours at her home environment, to confirm that the chosen size is appropriate for the user. Each usage will be followed by a vaginal examination. In case the investigator will determine that the subject should be fitted with a different size of the ProVATE device the subject will repeat this stage with a different device size until the suitable size is confirmed by the investigator.

Usage:

The subject will use the ProVATE device for at least 28 days during a 45 days period, at her home environment, and fill a usage diary. Each device will be used for at least 24 hours. At least one (1) follow-up phone call will be held with the subject per a week. After 14 usage days or following at least two (2) usages (the latest of them) the subject will be scheduled for vaginal examination at the clinic (visit four (4)).

End Of Use At the end of use the subject will return to the clinic (visit five (5)) for a vaginal examination and additional activities.

The following questionnaires will be filled at baseline and end of study: Quality Of Life (QoL) and POP symptoms. Satisfaction and Ease Of Use questionnaires will be filled at the end of use (visit 5) Up to four (4) ProVATE device models will be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 21-80 years
* Ability to use both hands and insert a device into the vagina
* Ability to attend the study site as explained by the investigator
* A symptomatic sensation of vaginal prolapse
* The subject has the ability to understand the nature of the study and sign the informed consent
* On examination, the presence of a vaginal wall prolapse of one or more sites
* On examination, POP-Q grade 2 - 4 POP is demonstrated
* A 61-91 mm pessary is well fitted
* A 61-91 mm pessary is well retained

Exclusion Criteria:

* Previous inability to accommodate with tampons or vaginal pessaries
* Subject is currently participating in another clinical study which may directly or indirectly affect the results of this study
* Co-morbid condition(s) or severe systemic disease that could limit the subject 's ability to participate in the study, or impact the scientific integrity of the study
* Subject is pregnant, or suspected to be pregnant or is planning to be pregnant during the course of the study
* Abnormal vaginal bleeding in the past 6 months
* Previous vaginal surgery during the last 3 months
* A severely atrophic vagina
* Existing vaginal or vulvar laceration
* Symptomatic vaginal infection as determined by physical examination and lab results
* Symptomatic urinary tract infection as determined by physical examination and lab results
* Recurrent urinary tract infections
* Abnormal cervical cytology

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Degree of prolapse and POP symptoms following ProVATE device insertion, compared to the degree of prolapse prior to the insertion of the ProVATE device (by vaginal examination) | At day 1 - baseline, and following at least 28 and up to 45 days of using the ProVATE vaginal pessary

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Site 01, Herzliya
  - Site 02, Herzliya
  - Site 03, Ramat HaSharon